CLINICAL TRIAL: NCT02401113
Title: Effect of Ursolic Acid of Loquat Extract on Function of Muscle in Human
Brief Title: Effect of Ursolic Acid of Loquat Extract on Function of Muscle
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, family medicine, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UrsolicAcid
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UA group (Experimental): UA group who takes Ursolic acid of Loquat Extract , 500 mg/ day during 12 weeks for treatment of muscle function improvement with relatively health adults
  Interventions: Dietary Supplement: UA group
- placebo group (Placebo Comparator): placebo group who takes a placebo, 500 mg/day for 12 weeks
  Interventions: Dietary Supplement: UA group

INTERVENTIONS:
Dietary Supplement: UA group — Ursolic Acid of Loquat Extract, 500mg/ day during 12 weeks

SUMMARY:
This randomized, placebo-controlled, double-blind study was designed to investigate the efficacy and tolerability of Ursolic Acid of Loquat Extract for treatment of muscle function improvement with relatively health adults. 54 subjects received 500 mg of Loquat Extract per day or a placebo for 12 weeks.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, double-blind study was designed to investigate the efficacy and tolerability of Ursolic Acid of Loquat Extract for treatment of muscle function improvement with relatively health adults. 54 subjects received 500 mg of Loquat Extract per day or a placebo for 12 weeks. Change over time in muscle fuction was evaluated by four outcomes: assessment of appendicular skeletal mass using DEXA (dual energy X-ray absorptiometry); quadriceps muscle power by Biodex; hand grib power; and Short Physical Performance Battery, SPPB.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-30KG/M2

Exclusion Criteria:

* > SERUM creatinine 1.2mg/dL
* > AST or ALT 60IU/L
* DM Patients

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
quadriceps muscle function | 12weeks

SECONDARY OUTCOMES:
ASM(appendicular skeletal mass) marker | 12weeks
Short Physical Performance Battery, SPPB | 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: SANG YEOUP Lee, Pf., Principal Investigator — Pusan National University Yangsan Hospital

REFERENCES:
- [Result] Prissadova N, Bozov P, Marinkov K, Badakov H, Kristev A. Effects of ursolic acid on contractile activity of gastric smooth muscles. Nat Prod Commun. 2015 Apr;10(4):565-6. PMID 25973477
- [Derived] Cho YH, Lee SY, Kim CM, Kim ND, Choe S, Lee CH, Shin JH. Effect of Loquat Leaf Extract on Muscle Strength, Muscle Mass, and Muscle Function in Healthy Adults: A Randomized, Double-Blinded, and Placebo-Controlled Trial. Evid Based Complement Alternat Med. 2016;2016:4301621. doi: 10.1155/2016/4301621. Epub 2016 Nov 24. PMID 27999607